CLINICAL TRIAL: NCT03444727
Title: Treatment Prior to Injection and Biopsy of the Vulva
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough enrollment
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Kirby Woodall, Resident Physician, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010101
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Vulvar Diseases; Anesthesia; Anesthesia, Local
Keywords: vulvar biopsy; ice; anesthesia; pain; vulva
MeSH Terms: conditions — Vulvar Diseases; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either pre-treatment with ice inside a sterile glove or with room-temperature water inside an exam glove.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice Pre-treatment (Experimental): Participants will hold an exam glove filled with ice to intended biopsy area for 30 seconds prior to preparation and local anesthetic injection.
  Interventions: Other: Ice Pre-treatment
- Room Temperature Water Pre-Treatment (Placebo Comparator): Participants will hold an exam glove filled with room temperature water to intended biopsy area for 30 seconds prior to preparation and local anesthetic injection.
  Interventions: Other: Room Temperature Water Pre-treatment

INTERVENTIONS:
Other: Ice Pre-treatment — Topical application of ice prior to local anesthetic injection.
  Arms: Ice Pre-treatment
Other: Room Temperature Water Pre-treatment — Topical application of room-temperature water prior to local anesthetic injection.
  Arms: Room Temperature Water Pre-Treatment

SUMMARY:
This study will compare pre-treatment with ice prior to injection of local anesthetic for vulvar biopsy to no pre-treatment and evaluate pain levels and patient satisfaction with the procedure.

DETAILED DESCRIPTION:
To diagnose skin conditions of the vulva and determine appropriate treatment, a biopsy is often taken as an outpatient procedure. Prior to biopsy, the skin is cleansed and injected with a numbing solution. These injections can be quite painful in this sensitive area.

Ice has been used as topical anesthesia in a number of sites, including the cornea, the skin, and particularly in the mouth prior to anesthetic injections. However, there is no evidence for using ice anesthesia prior to injections of the vulvar tissues.

The purpose of this study is to evaluate the efficacy of using ice as pre-treatment prior to the injection of local anesthetic for vulvar biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Undergoing vulva biopsy during clinic visit
* Willing and able to comply with study protocol
* Able to understand and provide informed consent

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Post-injection Pain Score | Immediately after local anesthetic injection
  Patient's self-reported visual analogue pain scale (100 millimeter) after injection of local anesthetic. Range from 0 to 100 mm, with 0 being least amount of pain and 100 being the most amount of pain.

SECONDARY OUTCOMES:
Post-procedure satisfaction score | Immediately after procedure
  Patient's self-reported visual analogue scale (100 millimeter) for satisfaction with the procedure. Range form 0mm to 100mm with 0 being the least satisfied and 100 being the most satisfied.
Post-procedure anxiety score | Immediately after procedure
  Patient's self-reported visual analogue scale (100 millimeter) score for anxiety level about having another vulvar biopsy in the future. Range from 0mm to 100mm, with 0 being the least anxious and 100 being the most anxious about a future procedure.
Post-procedure pain control score | Immediately after procedure
  Patient's self-reported visual analogue scale (100 millimeter) for satisfaction with pain control during procedure. Range from 0mm to 100mm with 0 being the least satisfied with pain control and 100mm being the most satisfied with pain control.
Post-biopsy pain score | Immediately after procedure.
  Patient's self-reports visual analogue pain scale (100 millimeter) score immediately after biopsy. Range from 0mm to 100mm, with 0 being the the least pain and 100 being the most pain.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Barnes, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Missouri Ob/Gyn Associated, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuwahara RT, Skinner RB. Emla versus ice as a topical anesthetic. Dermatol Surg. 2001 May;27(5):495-6. doi: 10.1046/j.1524-4725.2001.00343.x. PMID 11359502
- [Background] Chan HH, Lam LK, Wong DS, Wei WI. Role of skin cooling in improving patient tolerability of Q-switched Alexandrite (QS Alex) laser in nevus of Ota treatment. Lasers Surg Med. 2003;32(2):148-51. doi: 10.1002/lsm.10112. PMID 12561049
- [Background] Goel S, Chang B, Bhan K, El-Hindy N, Kolli S. "Cryoanalgesic preparation" before local anaesthetic injection for lid surgery. Orbit. 2006 Jun;25(2):107-10. doi: 10.1080/01676830600675392. PMID 16754218
- [Background] Leff DR, Nortley M, Dang V, Bhutiani RP. The effect of local cooling on pain perception during infiltration of local anaesthetic agents, a prospective randomised controlled trial. Anaesthesia. 2007 Jul;62(7):677-82. doi: 10.1111/j.1365-2044.2007.05056.x. PMID 17567343
- [Background] Dixit S, Lowe P, Fischer G, Lim A. Ice anaesthesia in procedural dermatology. Australas J Dermatol. 2013 Nov;54(4):273-6. doi: 10.1111/ajd.12057. Epub 2013 Apr 26. PMID 23617804
- [Background] Ghaderi F, Banakar S, Rostami S. Effect of pre-cooling injection site on pain perception in pediatric dentistry: "A randomized clinical trial". Dent Res J (Isfahan). 2013 Nov;10(6):790-4. PMID 24379869
- [Background] Lindsell LB, Miller DM, Brown JL. Use of topical ice for local anesthesia for intravitreal injections. JAMA Ophthalmol. 2014 Aug;132(8):1010-1. doi: 10.1001/jamaophthalmol.2014.1397. No abstract available. PMID 24945871
- [Background] Lathwal G, Pandit IK, Gugnani N, Gupta M. Efficacy of Different Precooling Agents and Topical Anesthetics on the Pain Perception during Intraoral Injection: A Comparative Clinical Study. Int J Clin Pediatr Dent. 2015 May-Aug;8(2):119-22. doi: 10.5005/jp-journals-10005-1296. Epub 2015 Aug 11. PMID 26379379
- [Background] Davoudi A, Rismanchian M, Akhavan A, Nosouhian S, Bajoghli F, Haghighat A, Arbabzadeh F, Samimi P, Fiez A, Shadmehr E, Tabari K, Jahadi S. A brief review on the efficacy of different possible and nonpharmacological techniques in eliminating discomfort of local anesthesia injection during dental procedures. Anesth Essays Res. 2016 Jan-Apr;10(1):13-6. doi: 10.4103/0259-1162.167846. PMID 26957683
- [Background] Bhadauria US, Dasar PL, Sandesh N, Mishra P, Godha S. Effect of injection site pre-cooling on pain perception in patients attending a dental camp at Life Line Express: a split mouth interventional study. Clujul Med. 2017;90(2):220-225. doi: 10.15386/cjmed-694. Epub 2017 Apr 25. PMID 28559708